CLINICAL TRIAL: NCT05303649
Title: Effects of Neuronavigated Theta Burst Stimulation in Therapy of Post-stroke Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Principal Investigator, Katarzyna Polanowska, Principal Investigator, Institute of Psychiatry and Neurology, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPiN_KP01
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Ischemic; Aphasia Non Fluent
Keywords: Aphasia; Stroke; Theta Burst Stimulation; Therapy; Rehabilitation; Noninvasive Transcranial Brain Stimulation
MeSH Terms: conditions — Ischemic Stroke; Aphasia, Broca; Aphasia; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermittent TBS (iTBS) of the left hemisphere plus behavioral aphasia therapy (Experimental): 15 sessions of 200-second of iTBS over the pars triangularis of Broca's area in the left hemisphere (BA 45), preceding 45-minutes of behavioral aphasia therapy.
  Interventions: Device: Noninvasive transcranial brain stimulation: excitatory iTBS; Behavioral: Individual speech-language therapy (SLT)
- Continuous TBS (cTBS) of the right hemisphere plus behavioral aphasia therapy (Experimental): 15 sessions of 40 seconds of cTBS over the pars triangularis of the right inferior frontal gyrus (BA 45 homologue), preceding 45-minutes of behavioral aphasia therapy.
  Interventions: Device: Noninvasive transcranial brain stimulation: inhibitory cTBS; Behavioral: Individual speech-language therapy (SLT)
- Sham TBS (sTBS) of the left hemisphere plus behavioral aphasia therapy (Sham Comparator): 15 sessions of sham TBS over the pars triangularis of Broca's area in the left hemisphere (BA 45), preceding 45-minutes of behavioral aphasia therapy.
  Interventions: Behavioral: Individual speech-language therapy (SLT); Device: Sham TBS simulating left hemispheric iTBS

INTERVENTIONS:
Device: Noninvasive transcranial brain stimulation: excitatory iTBS — 600 pulses (3 pulses at 50 Hz given every 200 milliseconds in 2-second trains at 10-second intervals, delivered at 80% of active motor threshold) generated by Magstim Super Rapid2 stimulator equipped with a figure-of-eight coil applied over BA 45 Device: Magstim Co., Wales, UK.
  Other Names: Magstim Super Rapid2
  Arms: Intermittent TBS (iTBS) of the left hemisphere plus behavioral aphasia therapy
Device: Noninvasive transcranial brain stimulation: inhibitory cTBS — 600 pulses (3 pulses at 50 Hz, repeated at 5 Hz, delivered at 80% of active motor threshold) generated by Magstim Super Rapid2 stimulator equipped with a figure-of-eight coil applied over BA 45 homologue Device: Magstim Co., Wales, UK.
  Other Names: Magstim Super Rapid2
  Arms: Continuous TBS (cTBS) of the right hemisphere plus behavioral aphasia therapy
Behavioral: Individual speech-language therapy (SLT) — 45 minutes training tailored to every patient's deficits, abilities and needs. Exercises used during each therapeutic session include: expressions tasks (naming and sentence building), complex utterances comprehension tasks, reading and writing exercises. Training is administered using paper-and-pencil tasks and computerized aphasia therapy program AfaSystem (Harpo sp.zoo, Poznań, Poland).
Device: Sham TBS simulating left hemispheric iTBS — Sham TMS coil positioned exactly like an active TMS coil resulting in a very good approximation of the auditory effects Device: Magstim Co., Wales, UK.
  Other Names: Magstim Super Rapid2
  Arms: Sham TBS (sTBS) of the left hemisphere plus behavioral aphasia therapy

SUMMARY:
Aphasia is an impairment in the ability to express and/or understand language, commonly observed after stroke to the language dominant (left) hemisphere. Despite natural tendency to spontaneous functional recovery in the first months post stroke and language improvement due to application of behavioral speech and language therapy (SLT), many aphasic patients do not achieve satisfactory level of verbal communication. The aim of the planned study is to explore the potential of the noninvasive repetitive Transcranial Magnetic Stimulation (rTMS) as a therapeutic tool for aphasia in addition to traditional behavioral therapy. In case of aphasia, studies on therapeutic effectiveness of rTMS aim to increase the activity of the language-dominant left cerebral hemisphere, which may be achieved in an indirect manner by inhibiting the activity of the opposite (right) hemisphere or in a direct manner by increasing the excitability of preserved language areas in the left hemisphere. In our study, we plan to administer the newest form of rTMS called Theta Burst Stimulation (TBS), which is safer than the conventional rTMS, even when used in the perilesional area. Computer-based neuronavigation system will be implemented to precisely localize stimulation targets, control administration of stimuli during rTMS sessions, and evaluate differences between participants regarding deviations from established stimulation points. 45 patients (all right-handed, polish native speakers, aged 18-75 years, diagnosed with non-fluent aphasia) will be enrolled in a randomized, double-blind, sham-controlled trial. Subjects will be randomly assigned to one of the three groups: 1) a group with excitatory intermittent TBS of the left hemisphere (iTBS group), 2) a group with inhibitory continuous TBS of the right hemisphere (cTBS group), 3) a group with sham TBS (sTBS group as a control group). Specific forms of stimulation will be carried out for three consecutive weeks (Monday to Friday; a total of 15 stimulation sessions). Immediately after each session of the stimulation, patients will undergo individual SLT. Assessment of language functioning will be carried out three times: before and after the therapy period, and 3 months after its completion. Results of the study will broaden knowledge about hemispherical mechanisms of language and speech recovery after stroke and provide insight into possibilities of their modulation for the purpose of post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* First-ever left middle cerebral artery ischemic stroke (brain damage localization confirmed by magnetic resonance imaging, MRI)
* 3 or more months from the onset of stroke
* Non-fluent aphasia (confirmed in the BDAE test) with functional communication difficulties ranging from mild to significant (grades from 2 to 4 in ASRS), marked difficulties in naming, and relatively preserved everyday speech comprehension
* Native Polish speaker
* Right-handedness prior to stroke
* Signing of the informed consent for the participation in the study.

Exclusion Criteria:

* Psychiatric and/or neurological comorbidity (e. g. dementia, depressive disorder, alcohol dependence)
* Diagnose of epilepsy or epileptic changes in EEG, also frequent losses of consciousness of unclear etiology which might suggest epileptic seizures
* History of any neurosurgical procedure around the head area
* 1.5 T MRI examination contraindications (metal elements in the body, e. g. implantable cardioverter-defibrillator, deep brain stimulation devices; claustrophobia)
* Regular intake of medication that could affect cortical excitability (e. g. antiepileptic or antipsychotic drugs, antidepressants, benzodiazepines) or medication influencing neuroplastic processes (e. g. dopamine)
* Significant cognitive impairment limiting patient's cooperation during assessment and behavioral aphasia therapy
* Visual deficits significantly hindering the perception of therapeutic tasks presented visually on a computer's screen
* New neurological episode (e. g. another brain stroke) or somatic illness (e. g. COVID-19) during the cycle of the therapy, requiring its interruption.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from pre-treatment assessment in the performance on a picture naming task | Pre-treatment assessment (within 2 days before starting the intervention), post-treatment assessment (within 2 days of completing the 15 days intervention)
  Total number of correctly named items (assessed: accuracy and speed of naming) from a set of 250 visually presented objects (200 noun names and 50 verb names; stimuli included in the set are diversified with regard to the articulation difficulty of corresponding words and their usage frequency in everyday speech).
Change from pre-treatment in the performance on the picture naming task at 3 months post-therapy (follow up assessment) | Pre-treatment and 3 months follow-up (post-treatment) assessment
  Total number of correctly named items from a set of 250 visually presented objects.
Change from post-treatment in the performance on the picture naming task at 3 months post-therapy | Post-treatment and 3 months follow-up assessment
  Total number of correctly named items from a set of 250 visually presented objects.
Change from pre-treatment assessment in the performance on a scene description task of three visually presented scenes | Pre-treatment assessment, post-treatment assessment (within 2 days of completing the 15 days intervention)
  (assessed: length and correctness of utterances).
Change from pre-treatment in the scene description task at 3 months post-therapy | Pre-treatment and 3 months follow-up
  Oral description of three visually presented scenes (assessed: length and correctness of utterances).
Change from post-treatment in the scene description task at 3 months post-therapy | Post-treatment and 3 months follow-up
  Oral description of three visually presented scenes (assessed: length and correctness of utterances).
Change from pre-treatment on the semantic fluency task | Pre-treatment and post-treatment (within 2 days of completing the 15 days intervention)
  Producing within a minute as many words as possible from 3 semantic categories: animals, fruit, clothes; assessed: total number of correctly generated items.
Change from pre-treatment on the semantic fluency task at 3 months post-therapy | Pre-treatment and 3 months follow-up
  Total number of correctly generated items such as animals, fruits, clothes.
Change from post-treatment on the semantic fluency task at 3 months post-therapy | Post-treatment and 3 months follow-up
  Total number of correctly generated items such as animals, fruits, clothes.

SECONDARY OUTCOMES:
Modified Communication Effectiveness Index (CETI) | Pre-treatment, post-treatment (within 2 days of completing the 15 day intervention) and on 3-month follow-up
  A questionnaire to complete by researcher and family member/caregiver. Contains descriptions of ten communication situations, patients' performance in each of them is assessed on a Likert-type scale (from 0 to 7). Higher score means better functional communication.

OTHER OUTCOMES:
The Polish version of short form of the Boston Diagnostic Aphasia Examination (BDAE) | Screening appointment (pre-enrollment assessment)
  Assesses the linguistic skills of adults with aphasia. This provides information for the diagnosis of the type of aphasia. Includes the six-point Goodglass and Kaplan's Aphasia Severity Rating Scale (ASRS; 0-5 points - lower score means more severe language impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna E Polanowska, PhD, Principal Investigator — Institute of Psychiatry and Neurology, Warsaw, Poland
Locations (1):
- Institute of Psychiatry and Neurology, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harvey DY, Mass JA, Shah-Basak PP, Wurzman R, Faseyitan O, Sacchetti DL, DeLoretta L, Hamilton RH. Continuous theta burst stimulation over right pars triangularis facilitates naming abilities in chronic post-stroke aphasia by enhancing phonological access. Brain Lang. 2019 May;192:25-34. doi: 10.1016/j.bandl.2019.02.005. Epub 2019 Mar 11. PMID 30870740
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A. Screening questionnaire before TMS: an update. Clin Neurophysiol. 2011 Aug;122(8):1686. doi: 10.1016/j.clinph.2010.12.037. Epub 2011 Jan 11. No abstract available. PMID 21227747
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Shah PP, Szaflarski JP, Allendorfer J, Hamilton RH. Induction of neuroplasticity and recovery in post-stroke aphasia by non-invasive brain stimulation. Front Hum Neurosci. 2013 Dec 24;7:888. doi: 10.3389/fnhum.2013.00888. PMID 24399952
- [Background] Schlaug G, Marchina S, Wan CY. The use of non-invasive brain stimulation techniques to facilitate recovery from post-stroke aphasia. Neuropsychol Rev. 2011 Sep;21(3):288-301. doi: 10.1007/s11065-011-9181-y. Epub 2011 Aug 14. PMID 21842404
- [Background] Szaflarski JP, Griffis J, Vannest J, Allendorfer JB, Nenert R, Amara AW, Sung V, Walker HC, Martin AN, Mark VW, Zhou X. A feasibility study of combined intermittent theta burst stimulation and modified constraint-induced aphasia therapy in chronic post-stroke aphasia. Restor Neurol Neurosci. 2018;36(4):503-518. doi: 10.3233/RNN-180812. PMID 29889086
- [Background] Szaflarski JP, Vannest J, Wu SW, DiFrancesco MW, Banks C, Gilbert DL. Excitatory repetitive transcranial magnetic stimulation induces improvements in chronic post-stroke aphasia. Med Sci Monit. 2011 Feb 25;17(3):CR132-9. doi: 10.12659/msm.881446. PMID 21358599
- [Background] Ball LJ, Beukelman DR, Pattee GL. Communication effectiveness of individuals with amyotrophic lateral sclerosis. J Commun Disord. 2004 May-Jun;37(3):197-215. doi: 10.1016/j.jcomdis.2003.09.002. PMID 15063143